CLINICAL TRIAL: NCT03362333
Title: Pain Neuroscience Education and Exercise Versus Exercise for University Students With Chronic Idiopathic Neck Pain: a Randomized, Controlled and Single Blind Study
Brief Title: Pain Neuroscience Education and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Dr, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCEDCSS-FMUP 18
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pain neuroscience education and exercise (Experimental): This group received pain neuroscience education and exercise once a week over 4 weeks
  Interventions: Other: Exercise; Other: Pain neuroscience education
- Exercise (Active Comparator): This group received exercise directed at the neck and shoulder regions once a week over 4 weeks
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercises were aimed at increasing the endurance and strength of the deep neck flexor and extensor muscles and of the scapular stabilizer muscles.
Other: Pain neuroscience education — Pain neuroscience education covered the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience.
  Arms: pain neuroscience education and exercise

SUMMARY:
This study examined the effects of pain neuroscience education plus exercise when compared with exercise only in university students with chronic idiopathic neck pain.

DETAILED DESCRIPTION:
This study examined the effects of pain neuroscience education plus exercise when compared with exercise only in university students with chronic idiopathic neck pain.

University students with chronic neck pain were randomly allocated to receive pain neuroscience education and exercise or exercise only and assessed at baseline, after the intervention and at 3 months follow up. Outcome variables were pain intensity (primary outcome), disability, fear of movement, catastrophizing, knowledge of pain neurophysiology, pressure pain thresholds and neck and scapular muscle endurance.

ELIGIBILITY:
Inclusion Criteria:

* Participants could enter the study if they had chronic idiopathic neck pain, defined as pain felt in the neck at least once a week in the previous 3 months and for which no cause had been established. Furthermore, they were required to have a minimum pain intensity in the previous week of 2 in the visual analogue scale.

Exclusion Criteria:

* Participants were excluded if they had had physiotherapy for their neck pain in the 6 months previous to the study, if they had rheumatic, nervous, cardiac and/or respiratory pathology that could prevent or make it difficult to do the exercises. Exclusion criteria were ascertained by self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | At the beginning
  Measured using the visual analogue scale
Pain intensity | 5 weeks
  Measured using the visual analogue scale
Pain intensity | At 3 months
  Measured using the visual analogue scale

SECONDARY OUTCOMES:
Deep neck flexor endurance | At the beginning
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Deep neck flexor endurance | 5 weeks
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Neck extensors endurance | At the beginning
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Neck extensors endurance | 5 weeks
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Scapular stabilizers endurance | At the beginning
  Method of assessment - physical test; Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
Scapular stabilizers endurance | 5 weeks
  Method of assessment - physical test; Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
Pressure pain thresholds | At the beginning
  Method of assessment - psychophysical test; Pressure was applied over the trapezius and at C5-C6 with a algometer until the participant first felt pain. The results was the quantity of force (in Kgf) supported by participants.
Pressure pain thresholds | 5 weeks
  Method of assessment - psychophysical test; Pressure was applied over the trapezius and at C5-C6 with a algometer until the participant first felt pain. The results was the quantity of force (in Kgf) supported by participants.
Disability | At the beginning
  Method of assessment - the neck pain disability index
Disability | 5 weeks
  Method of assessment - the neck pain disability index
Disability | 3 months
  Method of assessment - the neck pain disability index
catastrophizing | at beginning
  Method of assessment - Pain catastrophising scale
catastrophizing | 5 weeks
  Method of assessment - Pain catastrophising scale
catastrophizing | 3 months
  Method of assessment - Pain catastrophising scale
fear of movement | At the beginning
  method of assessment - the Tampa Scale
fear of movement | 5 weeks
  method of assessment - the Tampa Scale
fear of movement | 3 months
  method of assessment - the Tampa Scale
Knowledge of pain neurophysiology | at beginning
  method of assessment - scale; the neurophysiology of pain questionnaire
Knowledge of pain neurophysiology | 5 weeks
  method of assessment - scale; the neurophysiology of pain questionnaire
Knowledge of pain neurophysiology | 3 months
  method of assessment - scale; the neurophysiology of pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, PhD, Principal Investigator — University of Aveiro

IPD SHARING:
Plan to Share IPD: No